CLINICAL TRIAL: NCT00005068
Title: A Phase I Study of Oxaliplatin, CPT-11, 5-FU and Leucovorin in Patients With Solid Tumors
Brief Title: Combination Chemotherapy In Treating Patients With Metastatic or Unresectable Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Richard M. Goldberg, M.D., Mayo Clinic Cancer Center
Purpose: Treatment
Other Study IDs: CDR0000067673; U01CA069912 (NIH); P30CA015083 (NIH); 970109 (Other: Mayo Clinic Cancer Center)
Record Dates: First submitted 2000-04-06; First posted 2004-04-02 (Estimated); Last update posted 2011-08-03 (Estimated); Status verified 2011-08

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Fluorouracil; Irinotecan; Leucovorin; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: fluorouracil
Drug: irinotecan hydrochloride
Drug: leucovorin calcium
Drug: oxaliplatin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase I trial to determine the effectiveness of two different regimens of combination chemotherapy in treating patients who have metastatic or unresectable solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose of irinotecan, fluorouracil, and leucovorin calcium (Saltz regimen vs Mayo regimen) plus oxaliplatin (arm I vs arm II) in patients with metastatic or unresectable solid tumors. II. Determine the effect of irinotecan on the disposition of oxaliplatin in these patients. III. Assess the development of peripheral neuropathy in these patients on the Mayo regimen. IV. Determine the activity of these regimens in patients with metastatic solid tumors.

OUTLINE: This is a dose escalation study. Patients are entered to one of two treatment arms: Arm I (Saltz regimen): Patients receive irinotecan IV over 90 minutes, leucovorin calcium IV, and fluorouracil IV on days 1, 8, 15, and 22, followed by oxaliplatin IV over 2 hours on days 1 and 15. Courses repeat every 6 weeks. Arm II (Mayo regimen): Patients receive irinotecan IV over 90 minutes and oxaliplatin IV over 2 hours on day 1, followed by leucovorin calcium IV and fluorouracil IV over 90 minutes on days 2-5. Courses repeat every 3 weeks. Cohorts of 3-6 patients receive escalating doses of fluorouracil (one of two treatment doses for arm II), and one of two treatment doses of irinotecan and oxaliplatin until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose limiting toxicity. Patients are followed for 3 months.

PROJECTED ACCRUAL: Up to 60 patients will be accrued for this study within 8-14 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven metastatic or unresectable solid tumor for which no standard or curative therapy exists No CNS metastases

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: At least 12 weeks Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 times upper limit of normal (ULN) AST no greater than 5 times ULN Renal: Creatinine normal OR Creatinine clearance at least 60 mL/min Cardiovascular: No symptomatic congestive heart failure No unstable angina pectoris No cardiac arrhythmias No New York Heart Association class III or IV heart disease Neurologic: No peripheral neuropathy grade 2 or greater No uncontrolled seizure disorders Other: Not pregnant or nursing Fertile patients must use effective contraception No uncontrolled concurrent illness No active infection No history of allergy to platinum compounds, irinotecan, antiemetics, or antidiarrheals

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 4 weeks since prior immunotherapy At least 4 weeks since prior biologic therapy No concurrent immunotherapy Chemotherapy: At least 4 weeks since prior chemotherapy (6 weeks since nitrosoureas or mitomycin) and recovered No greater than 3 prior chemotherapy regimens for metastatic disease No other concurrent chemotherapy Endocrine therapy: Not specified Radiotherapy: No prior pelvic radiotherapy At least 4 weeks since other prior radiotherapy No prior radiotherapy to greater than 25% of bone marrow No concurrent radiotherapy Surgery: Not specified Other: No concurrent antiretroviral therapy for HIV positive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-01; Primary Completion 2003-06 (Actual); Study Completion 2003-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard M. Goldberg, MD, Study Chair — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Result] Goetz MP, Erlichman C, Windebank AJ, Reid JM, Sloan JA, Atherton P, Adjei AA, Rubin J, Pitot H, Galanis E, Ames MM, Goldberg RM. Phase I and pharmacokinetic study of two different schedules of oxaliplatin, irinotecan, Fluorouracil, and leucovorin in patients with solid tumors. J Clin Oncol. 2003 Oct 15;21(20):3761-9. doi: 10.1200/JCO.2003.01.238. Epub 2003 Sep 8. PMID 12963697